CLINICAL TRIAL: NCT00055003
Title: Effects of Hydrocortisone Infusion on Processing of Facially Expressed Emotion During Functional Magnetic Resonance Imaging
Brief Title: Effect of Hydrocortisone on the Brain
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030102; 03-M-0102
Record Dates: First submitted 2003-02-15; First posted 2003-02-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-18

CONDITIONS: Healthy
Keywords: Amygdala; Medial Prefrontal Cortex; Orbitofrontal Cortex; Cortisol; Memory; Glucocorticoid; Hydrocortisone; Stress; Perception; Affect; Healthy Volunteer; HV

SUMMARY:
The purpose of this study is to use brain imaging technology to examine the effect of the hormone hydrocortisone on the brain's response to various facial expressions.

Glucocorticoids can influence emotional behavior and cognition; when given long-term, the hormones may lead to mania or depression. One way glucocorticoids may influence emotional behavior is by affecting the activity of certain parts of the brain that participate in emotional processing. Brain imaging studies indicate that the amygdala, ventral medial prefrontal, and other prefrontal cortical areas of the brain are activated during tasks that require processing of emotional stimuli. These brain structures contain dense concentrations of glucocorticoid receptors. This study will use functional magnetic resonance imaging (fMRI) to study the brain activity of participants as they view faces that express different emotions. Participants will perform this task under a dose of either the glucocorticoid hydrocortisone or placebo (an inactive solution).

Participants in this study will be screened with a medical history, physical examination, blood tests, and an interview about their mood, degree of nervousness, and behavior. On Visit 1, participants will undergo screening and neuropsychological testing. For 3 days prior to Visit 2, participants will collect their saliva. During Visit 2, participants will undergo MRI scans of the brain after infusion with either a high or low dose of hydrocortisone or placebo. Participants will also undergo functional MRI (fMRI). Blood samples will be collected every 15 minutes during the scan. Following the MRI, participants will take attention and memory tests.

...

DETAILED DESCRIPTION:
Glucocorticoids influence performance on declarative memory tasks and tasks of memory for emotional information. The cognitive effects of exogenous glucocorticoids depend on dose, the time period between administration and testing, and the time of testing within the diurnal pattern of cortisol secretion. Additionally, glucocorticoid administration can influence mood, and with chronic administration glucocorticoids may lead to development of mania or depression.

A potential mechanism by which glucocorticoids may influence emotional behavior is via their effects on the neurophysiological activity of the amygdala and prefrontal cortical structures known to participate in emotional processing. Human imaging studies indicate that amygdala, ventral medial prefrontal, and other prefrontal cortical areas are activated during tasks requiring processing of affective stimuli. These data converge with lesion analysis and electrophysiological studies performed in humans or experimental animals to indicate that these structures participate in brain circuits that process emotional information. These brain structures contain dense concentrations of glucocorticoid and mineralocorticoid receptor mRNA, glucocorticoid receptors and mineralocorticoid receptors. Increased glucocorticoids appear to potentiate activation of the amygdala and affect processing of emotionally laden stimuli based on both experimental animal studies and correlational human studies.

The present study investigates the influence of glucocorticoids on the hemodynamic response that occurs while processing emotionally-valenced visual stimuli known to activate the amygdala and anatomically-related areas of the prefrontal cortex (PFC) in healthy humans. Functional magnetic resonance images will be acquired during the performance of tasks that involve viewing emotionally expressive faces both before and following either hydrocortisone (synthetic cortisol) (0.15 mg/kg or 0.45 mg/kg bolus) or placebo administration. The change in the BOLD signal in structures of interest will be compared across high dose cortisol, low dose cortisol and placebo conditions. In addition, the effects of hydrocortisone on relative blood flow in the amygdala and PFC will be assessed using an arterial spin labeling (ASL) technique to measure perfusion. The findings of this study will guide future research into the effects of glucocorticoids on emotional perception in subjects with mood disorders.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects will be between 18 and 50 years old.

Male and female subjects will be included.

Females will be studied in the luteal phase.

All subjects must be able to give written informed consent prior to participation in this study.

EXCLUSION CRITERIA:

Children less than 18.

Individuals with any major medical or neurological disorder, or taking any medication within 3 weeks of scanning that is likely to influence CBF or metabolism, or having any endocrine condition expected to be associated with abnormal HPA axis function.

Individuals who meet DSM-IV criteria for alcohol and/or substance abuse within 1 year prior to screening or lifetime history of substance dependence.

Individuals with a current or past history of other axis I psychiatric disorders.

Individuals with first-degree family members with current or past history of mood disorder.

Women of childbearing potential who have a positive pregnancy test who are currently nursing.

Individuals who have experienced serious suicidal ideation or attempt within the past 6 months.

Smokers are ineligible to participate.

Women with irregular menstrual cycles or taking oral contraceptives.

Those with a weight greater than 100 kgs.

Those with previous allergic reactions or hypersensitivity to hydrocortisone.

General exclusions for MRI imaging, such as having had a cardiac pacemaker or ferromagnetic object implanted through surgical intervention or accident, e.g. shrapnel.

Those with a history of peptic ulcer disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2003-02-13; Study Completion 2010-11-18

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Buchanan TW, Lovallo WR. Enhanced memory for emotional material following stress-level cortisol treatment in humans. Psychoneuroendocrinology. 2001 Apr;26(3):307-17. doi: 10.1016/s0306-4530(00)00058-5. PMID 11166493
- [Background] Nejtek VA. High and low emotion events influence emotional stress perceptions and are associated with salivary cortisol response changes in a consecutive stress paradigm. Psychoneuroendocrinology. 2002 Apr;27(3):337-52. doi: 10.1016/s0306-4530(01)00055-5. PMID 11818170
- [Background] Newcomer JW, Selke G, Melson AK, Hershey T, Craft S, Richards K, Alderson AL. Decreased memory performance in healthy humans induced by stress-level cortisol treatment. Arch Gen Psychiatry. 1999 Jun;56(6):527-33. doi: 10.1001/archpsyc.56.6.527. PMID 10359467